CLINICAL TRIAL: NCT03684473
Title: An Online CBT, Mindfulness Meditation, and Trauma-informed Yoga Intervention (CBT-MY) for Young Adults With Posttraumatic Stress Disorder: Evaluating Psychometric and Psychophysiology Outcomes
Brief Title: An Online CBT, Mindfulness Meditation & Yoga (CBT-MY) Intervention for Posttraumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: York University (Other)
Responsible Party: Principal Investigator, Paul Ritvo, Professor & Clinical Psychologist, York University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-208
Record Dates: First submitted 2018-08-09; First posted 2018-09-25 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Posttraumatic Stress Disorders; PTSD
Keywords: Yoga; Mindfulness Meditation; Online; Posttraumatic Stress Disorder; Young Adulthood
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yoga Intervention (Experimental): Participants in the intervention condition will be assigned to an 8-week online delivered trauma-informed yoga protocol focused on home-based daily practice of yoga and mindfulness meditation.
  Interventions: Behavioral: Online Mindfulness-Based CBT & Trauma-Informed Yoga Intervention

INTERVENTIONS:
Behavioral: Online Mindfulness-Based CBT & Trauma-Informed Yoga Intervention — 8 Weekly Online modules consisting of one weekly video of yoga postures combined with breath awareness and daily guided meditation audios, and a breath technique manual form the foundation of the intervention. The trauma-informed component of the program uses specific language, movement cues, teacher qualities, and physical assists. The yoga intervention will emphasize full choice and control of the participant through invitational language such as, "when you are ready", "if you like" before each body posture cue. Based on trauma-informed yoga best practices, a predictable foundation of yoga postures (with variations) will be followed in a consistent order each session to allow participants to anchor to the series.
  Other Names: Online Trauma-Informed Mindfulness-Based CBT Intervention

SUMMARY:
Post-traumatic stress disorder (PTSD), a chronic, debilitating condition, is a growing public health concern as the Canadian population has the highest PTSD prevalence worldwide (9.2%; 3.7 million people). PTSD is linked with other comorbid mental health disorders (e.g., depression) and increased risk of chronic disease (e.g., cardiovascular disease, obesity) which presents challenges as far as selection of the appropriate treatment approach. Adjunctive treatment approaches for PTSD that include somatic-sensory body awareness (e.g., mindfulness, yoga) have been shown to be viable treatment options to reduce stress-related symptoms and enhance emotion regulation. Online treatment delivery for mental health disorders demonstrate similar reductions in self-reported symptoms as face-to-face methods and emphasize accessibility, reduced costs, and enhanced appeal to certain demographic groups. A target population at risk of untreated PTSD symptoms that may benefit from an online treatment is young adults, 18-34 yrs., who have experienced childhood trauma. No known clinical trial (CT) has addressed the effectiveness of a brief (8-week) online trauma-informed yoga intervention using both self-report and objective psychophysiology measures. The purpose of this study is to evaluate changes in self-reported PTSD symptoms and objectively measured biomarkers of autonomic regulation via pupil dilation and heart-rate-variability (HRV) following an 8-week single-arm experimental design. It is hypothesized that clinically significant reductions of: 1) PTSD total symptom severity by 10% and 2) significant reductions in pupil dilation at post-intervention and; 3) significant increases in HRV at post-intervention. This is the first study to examine objective markers of autonomic regulation among an at-risk population using multiple novel technologies (e.g., Eye Tracking Glasses, HRV) and comparing two theoretically-linked measures (e.g., HRV, Pupillometry). Comparisons of psychophysiology data with a cross-sectional convenience sample with no history of clinical PTSD or mental health conditions were made.

DETAILED DESCRIPTION:
Post-traumatic stress disorder (PTSD), a chronic, debilitating condition, is a growing public health concern as the Canadian population has the highest PTSD prevalence worldwide (9.2%; 3.7 million people). PTSD is linked with several co-morbid mental health disorders (e.g., depression) and increased risk of chronic disease (e.g., cardiovascular disease, obesity) which presents challenges as far as the determination of appropriate treatment. Adjunctive treatment approaches for PTSD that include somatic-sensory body awareness (e.g., mindfulness, yoga) have been shown to be viable treatment options to reduce stress-related symptoms and enhance emotion regulation. Online treatment deliveries for mental health disorders demonstrate similar reductions in self-reported symptoms as face-to-face methods and emphasize accessibility, reduced costs, and enhanced appeal to certain demographic groups. A target population at risk of untreated PTSD symptoms that may benefit from an online treatment is young adults, 18-34 yrs., who have experienced trauma during pre-adult development. No known clinical trial (CT) has addressed the effectiveness of a brief (8-week) online trauma-informed yoga intervention using both self-report and objective psychophysiology measures. This study evaluates such an intervention in terms of changes in self-reported PTSD symptoms and objectively measured biomarkers of autonomic regulation via pupil dilation and heart-rate-variability (HRV) following an 8-week single-arm experimental design. It is hypothesized that results will demonstrate clinically significant reductions of: 1) PTSD total symptom severity; 2) statistically significant reductions in pupil dilation and; 3) significant increases in HRV at post-intervention. This is the first study to examine objective markers of autonomic regulation in an at-risk population using multiple novel technologies (e.g., Eye Tracking Glasses, HRV) that compare two theoretically-linked measures (e.g., HRV, Pupillometry). Comparisons of psychophysiology data with a cross-sectional convenience sample with no history of clinical PTSD or mental health conditions are made

ELIGIBILITY:
Inclusion Criteria:

* Exposure to 1+ Lifetime Traumatic Events (LEC-5)
* Met clinical PTSD criteria and a minimum PTSD score of ≥ 12 on the Clinician Administered Posttraumatic Stress Scale (CAPS-5)
* 18-34 years of age

Exclusion Criteria:

* current/ongoing trauma (e.g., current physical or sexual abuse) within the last month
* current unstable medical condition
* current active suicide risk/self-harm and/or drug addiction
* current pregnancy/breastfeeding
* current yoga attendance within the last month
* no access to the internet

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Posttraumatic Stress Symptoms on the Clinician Administered Posttraumatic Stress Scale for the Diagnostic and Statistical Manual of Mental Disorders (CAPS-5) | Baseline and 8-weeks
  A 30-item structured in-person interview with a trained clinician to confirm a current diagnosis of PTSD and associated symptoms based on a single index traumatic event (e.g., most recent, most severe). A single severity/distress score is calculated based on the frequency and intensity of a symptom using a 5-point scale (0 = absent/ no symptom; 1 = Mild/Symptom minimal; 2 = Moderate/Symptom Clearly Present; 3 = Severe/Symptom Pronounced; 4 = Extreme/Symptom is extreme/incapacitating). For a clinically significant symptom to be deemed present, a minimum frequency of twice per month or "some of the time" (approximately 20-30%) plus a minimum intensity of "clearly present" must be reported. Scores range from 0 to 80.

SECONDARY OUTCOMES:
Change in Heart Rate Variability | Baseline and 8-weeks
  Participants will undergo a 5-minute neutral stimulus, 5-minute emotional stimulus task, and 10-minute guided meditation protocol. Electrocardiogram (ECG) recordings will be collected using a 4-channel data acquisition system, which uses 2 adhesive electrodes applied to the chest and a ground electrode on the ankle. Frequency-based metrics represent respiratory-based modulation of the autonomic nervous system (ANS). The primary three spectral components for ECG recordings are very low frequency (VLF; 0.003-0.04 Hz), low frequency (LF; 0.04-0.15 Hz), and high frequency (HF; 0.15-0.4 Hz). Greater power in the HF band is considered to reflect respiratory sinus arrhythmia as it reflects HR variation attributed to parasympathetic (vagal) tone. Additionally, a ratio of LF to HF power will provide a marker of ANS regulation in all participants. A higher LF-HF ratio indicates "sympathetic dominance", whereas values closer to 0 reflect ANS balance.
Change in Pupil Diameter | Baseline and 8-weeks
  Participants will wear specialised eye tracking glasses to obtain pupil dilation recordings. Accordingly, participants will be presented with a plain, neutral stimulus and asked to focus their eyes on a fixation cross on the computer. Baseline (BL) pupil diameter will be captured in the 500ms directly preceding the emotional stimulus. Participants will undergo an emotional stimulus (ES) task viewing standardized emotional images (e.g., happy, sad) on a computer screen followed by a guided 10-minute meditation (GM) phase. Average peak stimulus pupil dilation will be calculated during each phase (BL, ES, GM). Increased pupil dilation reflects sympathetic nervous system dominance.
Change in Respiration Rate | Baseline and 8-weeks
  Participants will undergo a 5-minute neutral stimulus, 5-minute emotional stimulus task, and 10-minute guided meditation protocol. A respiratory belt transducer will be worn around the abdomen at the same time heart rate and pupil diameter are being measured. The respiratory belt transducer is measures changes in chest diameter resulting from breathing by producing a linear voltage proportional to changes in length and connects directly to a Pod (DIN) Port on the electrocardiogram machine. Breaths will be measured and recorded as the number of breaths per minute.

OTHER OUTCOMES:
Change in Posttraumatic Stress Disorder Checklist for Diagnostic and Statistical Manual of Mental Disorders - Civilian Version (PCL-5) | Baseline and 8-weeks
  The PCL-5 is a standardised 20-item self-report scale for PTSD symptoms. Participants indicate how much they have been bothered by a symptom item listed over the past month using a five-point Likert scale ranging from 0 = Not at all to 4 = Extremely. The PCL-5 is easily scored by summing all of the items for a total symptom severity score ranging between 0 to 80. Clinically meaningful PTSD symptoms are present if items are rated as a minimum of 2 = "Moderately" or higher.
Change in Beck Anxiety Inventory (BAI) | Baseline and 8-weeks
  The BAI is a 21-item self-report inventory to assess symptoms of anxiety within the last two weeks. Respondents rate how much each of the 21 symptoms bothered them in the past month on a four-point ordinal Likert scale from 0 = "not at all" to 3 = "severely, it bothered me a lot". Scoring for the BAI ranges from a minimum of 0 to a maximum of 63 based on summing the scores for all items. The following empirically supported cutoffs are followed for the interpretation of scores: 0-9 = normal/no anxiety, 10-18 = mild to moderate anxiety, 19-29 = moderate to severe anxiety, 30-63 = severe anxiety.
Change in Beck Depression Index-II (BDI-II) | Baseline and 8-weeks
  Depression symptoms will be assessed using the BDI-II, a 21-item self-report survey. The BDI-II evaluates symptoms and attitudes related to depression using a four-level weighted Likert response scale ranging from 0 = not present to 3= severe. The participant is instructed to respond to items pertaining to how they were feeling in the past two weeks. Scoring for the BDI-II ranges from 0 to a maximum score of 63; empirically informed cutoff scores for severity of depression include the following: 0-13 = minimal, 14-19 = mild, 20-28 = moderate, 29-63 = severe.
Change in Five Facet Mindfulness Questionnaire (FFMQ) | Baseline and 8-weeks
  Daily Mindfulness will be measured using the 39-item FFMQ. The FFMQ assesses changes in mindfulness tendencies (e.g., non-judgement of inner experience) before and after a mindfulness-based intervention. The FFMQ measures five mindfulness-based factors including non-reactivity, observing, describing, non-judgement, and acting with awareness. Item scores range on a five-level Likert scale of 1 = never or rarely true to 5 = very often or always true. The FFMQ is scored by summing all item responses and total scores range from 0 to 195, with higher scores indicating greater levels of mindfulness.
Change in Pain Catastrophizing Scale (PCS) | Baseline and 8-Weeks
  Catastrophic thinking in relation to bodily pain will be measured using the 13-item self-report Pain Catastrophizing Scale. The PCS is a self-report measure, consisting of 13 items scored from 0 to 4, resulting in a total possible score of 52. The higher the score, the more catastrophizing thoughts are present. Previous studies have shown a cutoff of more than 30 points to be associated with clinical relevance. This measure has been found to have good psychometric properties, including high test-retest reliability and high internal consistency (Chronbach's alpha = 0.87-0.95). Some examples of the items include: "I keep thinking about how badly I want the pain to stop; I worry all the time about whether the pain will end; and I become afraid that the pain may get worse."
24-Hour Recall of Pain using the Brief Pain Inventory - Short Form (BPI) | Baseline and 8-Weeks
  The Brief Pain Inventory - Short Form is a 9 item self-administered questionnaire used to evaluate the severity of a participant's pain and the impact of this pain on their daily functioning. The patient is asked to rate their worst, least, average, and current pain intensity, list current treatments and their perceived effectiveness, and rate the degree that pain interferes with general activity, mood, walking ability, normal work, relations with other persons, sleep, and enjoyment of life on a 10 point scale. The assessment produces a mean pain severity score and mean pain interference score. Higher scores indicate greater pain severity and interference.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Ritvo, PhD, Study Director — York University, Toronto, Ontario, Canada
Locations (1):
- York University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kirk MA, Taha B, Dang K, McCague H, Hatzinakos D, Katz J, Ritvo P. A Web-Based Cognitive Behavioral Therapy, Mindfulness Meditation, and Yoga Intervention for Posttraumatic Stress Disorder: Single-Arm Experimental Clinical Trial. JMIR Ment Health. 2022 Feb 28;9(2):e26479. doi: 10.2196/26479. PMID 34499613